CLINICAL TRIAL: NCT06004544
Title: Prospective Pakistan Registry of Echocardiographic Screening in Asymptomatic Pregnant Women
Acronym: PRESAP
Status: Recruiting | Type: Observational
Sponsor: National Institute of Cardiovascular Diseases, Pakistan (Other)
Collaborators: Jinnah Postgraduate Medical Centre (Other Government)
Responsible Party: Principal Investigator, Sabha Bhatti, Professor, National Institute of Cardiovascular Diseases, Pakistan
Other Study IDs: IRB-33/2023
Record Dates: First submitted 2023-08-06; First posted 2023-08-22 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Cardiovascular Diseases in Pregnancy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Consecutive obstetric patients attending routine antenatal visits were enrolled in this ongoing registry. A standardized 2D transthoracic echocardiogram (TTE) protocol was employed. Ejection fraction (EF) was quantified using biplane Simpson's method.

DETAILED DESCRIPTION:
Consecutive obstetric patients attending routine antenatal visits were enrolled in this ongoing registry. A standardized 2D transthoracic echocardiogram (TTE) protocol was employed, including parasternal long and short, apical 4- and 2-chamber views. Continuous wave and pulse wave Doppler were used to assess left ventricular outflow tract (LVOT) gradients. Left ventricular (LV) function was quantified using biplane Simpson's method and visually assessed by two independent readers. Patients with significant valve disease or congenital heart disease underwent complete TTE. Those diagnosed with LV dysfunction or other cardiovascular diseases (CVD) were referred to the Cardio-Obstetrics clinic for further management and long-term follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Obstetric patients attending routine antenatal visits

Exclusion Criteria:

* Patients refused to give consent for echocardiography or participation in the study

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Consecutive obstetric patients attending routine antenatal visits
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2023-02-06 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants found to have abnormal left ventricular function | At the time of screening echocardiogram
  Prevalence of Left ventricular dysfunction (Ejection Fraction<55%)
Number of participants found to have abnormal heart valve function | At the time of screening echocardiogram
  Structural heart abnormalities (valvular heart lesions classified as mild, moderate and severe)

SECONDARY OUTCOMES:
Number of participants found to have adverse Maternal outcomes | At the time of delivery
  Maternal Mortality, Cardiogenic shock
Number of participants found to have adverse Fetal outcomes | At the time of delivery
  Infant Mortality, Infant birth weight (kg)

CONTACTS AND LOCATIONS:
Overall Officials: Sabha Bhatti, MD, Principal Investigator — National Institute of Cardiovascular Diseases
Locations (1):
- National Institute of Cardiovascular Diseases (NICVD), Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bhatti S, Naz S, Gurmani S, Yasmin H, Atif U, Karim M, Ahmed S, Zehra K, Hakeem A, Qamar N. Prospective Pakistan Registry of Echocardiographic Screening in Asymptomatic Pregnant Women. JACC Adv. 2024 Sep 2;3(12):101215. doi: 10.1016/j.jacadv.2024.101215. eCollection 2024 Dec. PMID 39817089